CLINICAL TRIAL: NCT03792061
Title: Adopting Strategy Training to Improve Participation Performance of Individuals With Cognitive Impairments After Stroke
Brief Title: Enhancing Community Participation for Stroke Survivors With Cognitive Impairments
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Feng-Hang Chang, Associate Professor, Graduate Institute of Injury Prevention and Control, Taipei Medical University, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201804055
Record Dates: First submitted 2019-01-01; First posted 2019-01-03 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Cognitive Impairment
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy Training (Experimental): Strategy training is an activity intervention training approach developed based on the theoretical tenets of metacognitive training. The purpose of strategy training is to guide individuals to generate problem-solving skills to address challenges that they identify in daily activities.
  Interventions: Behavioral: Strategy Training
- Reflective listening (No Intervention): Participants in the control group will receive dose-matched non-active intervention carried out by a trained research staff. The staff will use scripted questions to provoke participants to describe their experiences and feelings about their disease and their usual-care rehabilitation activities.

INTERVENTIONS:
Behavioral: Strategy Training — This approach is different from traditional direct skill training, which emphasizes clinicians' responsibility on identifying their patients' challenges in performing activities and teaching patients task-specific problem-solving strategies. Strategy training, on the other hand, requires clinicians to take a role as a facilitator, guiding participants to learn through prompts and questions. In the training process, participants learn to develop their own problem-solving strategies and work through the problems they have, through which they can develop self-efficacy and confidence to manage participation challenges. Participants can also generalize the strategies they learn to other similar problems they encounter in daily life.
  Arms: Strategy Training

SUMMARY:
Abstract

Method: Participants with a diagnosis of stroke and have cognitive impairment (a score of 3 or more on the Executive Interview, 14-item version) will be randomly assigned to the intervention group and the attention control group at a 1:1 ratio. Each session will be around 45 minutes and will be delivered 1 to 2 sessions per week for 12 to 15 sessions.

Outcome measures including the Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D), Canadian Occupational Performance Measure(COPM), Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms, Wisconsin Card Sorting Task (WCST), Stroop Test, Montreal Cognitive Assessment (MoCA), Trail-Making Test (TMT A and B), The National Institutes of Health Stroke scale (NIHSS), modified Rankin Scale (MRS), Euro-QoL-5-Dimension (EQ-5D) and Participation Strategies Self Efficacy Scale (PS-SES) will be administered at baseline (T1), post-intervention (T2), 3-month follow-up (T3), 6-month follow-up (T4), and 12-month follow-up (T5).

Of the recruited participants, 50 will recieve the fMRI tests (including the resting-state scan, the fMRI scan with Stroop Test and TMT tasks, and the anatomical structure scan) at baseline, post-intervention, and 6month follow-up.Data will be analyzed using multiple linear regression models and mixed-effects regression models.

DETAILED DESCRIPTION:
The proposed study will examine the efficacy of a newly developed intervention program, the Optimizing Participation after Stroke through Strategy-training (OPASS) program on improving participation in productivity, social activities, and community among community-dwelling people with cognitive impairments after stroke. The OPASS program were developed based on the theoretical tenets of strategy training, with the goal of helping participants to set their participation goals, identify barriers to their performance, develop strategies to address these barriers, and generalize their learning through iterative practice. To examine the efficacy of OPASS, the following objectives will be addressed in this study:

1. To examine whether, compared to a control group, participating in the OPASS program will improve participation in productivity, social, and community domains in stroke survivors with cognitive impairments;
2. To determine whether the changes in participation after the intervention is correlated with changes in applied cognition, daily activities, executive functioning, and self-efficacy.
3. To examine whether the intervention effect sustains at 3-, 6-, and 12-month following the intervention.

To address this purpose, parallel-group randomized controlled trial will be implemented to assess the efficacy of the OPASS program in comparison to the control group. An expected sample of 210 adults with stroke-related cognitive impairments and are undergoing outpatient rehabilitation services will be recruited from our collaborative sites in Northern Taiwan. These participants will be randomly assigned to the intervention group and the attention control group at a 1:1 ratio.

Outcome measures including the Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D), Canadian Occupational Performance Measure(COPM), Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms, Wisconsin Card Sorting Task (WCST), Stroop Test, Montreal Cognitive Assessment (MoCA), Trail-Making Test (TMT A and B), The National Institutes of Health Stroke scale (NIHSS), modified Rankin Scale (MRS), Euro-QoL-5-Dimension (EQ-5D) and Participation Strategies Self Efficacy Scale (PS-SES) will be administered at baseline (T1), post-intervention (T2), 3-month follow-up (T3), 6-month follow-up (T4), and 12-month follow-up (T5). Data will be analyzed using multiple linear regression models and mixed-effects regression models. Of the recruited participants, 100 will recieve the fMRI tests (including the resting-state scan, the fMRI scan with Stroop Test and TMT tasks, and the anatomical structure scan) at baseline(T1), post-intervention(T2), and 12-month follow-up (T5). Data will be analyzed using multiple linear regression models and mixed-effects regression models.

Qualitative in-depth interviews with participants, caregivers, and therapists will be conducted following the intervention. Data regarding the interviewees' experiences, satisfaction, and their perceived effectiveness of the intervention will be collected. Transcribed data will be coded by two independent coders and analyzed with thematic analysis method.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20 years and older
* Has a diagnosis of stroke
* Understand Mandarin
* Has cognitive impairment (a score of 3 or more on the Executive Interview, 14-item version)
* Provide informed consent

Exclusion Criteria:

* Have severe aphasia
* Have a pre-stroke diagnosis of dementia, current major depressive disorder, substance use, or other psychiatric disorders that may impede them from continually participating in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-01-13 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | From baseline to 6-8 weeks (post-intervention)
  The PM-3D4D is a 24-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community.

SECONDARY OUTCOMES:
Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms | From baseline to up to 6-8 weeks (post-intervention)
  The AM-PAC consists of three subscales that assesses three activity domains: basic mobility (18 items), daily activity (15 items), and applied cognitive (19 items). Each item asks the respondent to rate the difficulty to perform specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms | From baseline to 3-month follow-up
  The AM-PAC consists of three subscales that assesses three activity domains: basic mobility (18 items), daily activity (15 items), and applied cognitive (19 items). Each item asks the respondent to rate the difficulty to perform specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms | From baseline to 6-month follow-up
  The AM-PAC consists of three subscales that assesses three activity domains: basic mobility (18 items), daily activity (15 items), and applied cognitive (19 items). Each item asks the respondent to rate the difficulty to perform specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care (AMPAC) Outpatient Short Forms | From baseline to 12-month follow-up
  The AM-PAC consists of three subscales that assesses three activity domains: basic mobility (18 items), daily activity (15 items), and applied cognitive (19 items). Each item asks the respondent to rate the difficulty to perform specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
HEAL positive outlook questionnaire | From baseline to up to 6-8 weeks (post-intervention)
  he HEAL positive outlook questionnaire will be used to assess participant's positive attitude.
General self-efficacy Scale (GSES) | From baseline to up to 6-8 weeks (post-intervention)
  The GSES was developed to measure self-efficacy in managing home participation, community participation, productivity, communication, staying organized, and advocating for resources. The scale consists of 35 items. Each item is rated using a 1-10 Likert scale, with higher score indicating greater self-efficacy.
General self-efficacy Scale (GSES) | From baseline to 3-month follow-up
  The GSES was developed to measure self-efficacy in managing home participation, community participation, productivity, communication, staying organized, and advocating for resources. The scale consists of 35 items. Each item is rated using a 1-10 Likert scale, with higher score indicating greater self-efficacy.
General self-efficacy Scale (GSES) | From baseline to 6-month follow-up
  The GSES was developed to measure self-efficacy in managing home participation, community participation, productivity, communication, staying organized, and advocating for resources. The scale consists of 35 items. Each item is rated using a 1-10 Likert scale, with higher score indicating greater self-efficacy.
General self-efficacy Scale (GSES) | From baseline to 12-month follow-up
  The GSES was developed to measure self-efficacy in managing home participation, community participation, productivity, communication, staying organized, and advocating for resources. The scale consists of 35 items. Each item is rated using a 1-10 Likert scale, with higher score indicating greater self-efficacy.
Canadian Occupational Performance Measure (COPM) | From the first session to the last session of the study, up to 8 weeks
  The COPM inquires the client to identify important goals in their daily life and rate their performance and satisfaction for each goal on a 10-point visual analog scale.
Stroop Test | From baseline to up to 6-8 weeks (post-intervention)
  Participants will be asked to read out the ink color of the word as accurately and as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded. Construct validity of the Stroop Test in the TBI population has been published.
Stroop Test | From baseline to 3-month follow-up
  Participants will be asked to read out the ink color of the word as accurately and as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded. Construct validity of the Stroop Test in the TBI population has been published.
Stroop Test | From baseline to 6-month follow-up
  Participants will be asked to read out the ink color of the word as accurately and as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded. Construct validity of the Stroop Test in the TBI population has been published.
Stroop Test | From baseline to 12-month follow-up
  Participants will be asked to read out the ink color of the word as accurately and as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded. Construct validity of the Stroop Test in the TBI population has been published.
Trail-Making Test (TMT A and B) | From baseline to up to 6-8 weeks (post-intervention)
  Trail-Making Test (TMT A and B) will be used to measure sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in an ascending order (1-A-2-B-3-C...). The Time to complete TMT A and B will be calculated, in which a longer completion time will indicate poorer outcome. This instrument was validated in healthy people, patients with head injury, vascular disorders, and other diverse populations.
Trail-Making Test (TMT A and B) | From baseline to 3-month follow-up
  Trail-Making Test (TMT A and B) will be used to measure sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in an ascending order (1-A-2-B-3-C...). The Time to complete TMT A and B will be calculated, in which a longer completion time will indicate poorer outcome. This instrument was validated in healthy people, patients with head injury, vascular disorders, and other diverse populations.
Trail-Making Test (TMT A and B) | From baseline to 6-month follow-up
  Trail-Making Test (TMT A and B) will be used to measure sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in an ascending order (1-A-2-B-3-C...). The Time to complete TMT A and B will be calculated, in which a longer completion time will indicate poorer outcome. This instrument was validated in healthy people, patients with head injury, vascular disorders, and other diverse populations.
Trail-Making Test (TMT A and B) | From baseline to 12-month follow-up
  Trail-Making Test (TMT A and B) will be used to measure sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in an ascending order (1-A-2-B-3-C...). The Time to complete TMT A and B will be calculated, in which a longer completion time will indicate poorer outcome. This instrument was validated in healthy people, patients with head injury, vascular disorders, and other diverse populations.
Montreal Cognitive Assessment (MoCA) | From baseline to up to 6-8 weeks (post-intervention)
  MoCA Test allows people to quickly assess a patients cognitive health.
Montreal Cognitive Assessment (MoCA) | From baseline to 3-month follow-up
  MoCA Test allows people to quickly assess a patients cognitive health.
Montreal Cognitive Assessment (MoCA) | From baseline to 6-month follow-up
  MoCA Test allows people to quickly assess a patients cognitive health.
Montreal Cognitive Assessment (MoCA) | From baseline to 12-month follow-up
  MoCA Test allows people to quickly assess a patients cognitive health.
The National Institutes of Health Stroke scale (NIHSS) | From baseline to 3-month, 6-month, and 12-month follow-ups
  The National Institutes of Health Stroke scale (NIHSS) will be used to assess participant's health related quality of life.
modified Rankin Scale (MRS) | From baseline to 3-month, 6-month, and 12-month follow-ups
  The modified Rankin Scale (MRS) will be used to assess participant's health related quality of life.
Euro-QoL-5-Dimension (EQ-5D) | From baseline to 3-month, 6-month, and 12-month follow-ups
  The Euro-QoL-5-Dimension (EQ-5D) will be used to assess participant's health related quality of life.
Qualitative data | After intervention, an average of 2 months
  Qualitative in-depth interviews with participants, caregivers, and therapists will be conducted following the intervention. Data regarding the interviewees' experiences, satisfaction, and their perceived effectiveness of the intervention will be collected.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | From baseline to 3-month follow-up
  The PM-3D4D is a 24-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | From baseline to 6-month follow-up
  The PM-3D4D is a 24-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | From baseline to 12-month follow-up
  The PM-3D4D is a 24-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Hang Chang, ScD, Principal Investigator — Taipei Medical University
Locations (4):
- Taiwan (4):
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
The IPD is not planned to be shared.

REFERENCES:
- [Derived] Hsu SP, Hung TH, Lin YN, Kang JH, Han DS, Chiu V, Liou TH, Wu YH, Ni PS, Skidmore ER, Chang FH. Enhancing Societal Participation for Stroke Survivors With Cognitive Impairments: A Randomized Controlled Trial. J Am Heart Assoc. 2025 Oct 7;14(19):e042295. doi: 10.1161/JAHA.125.042295. Epub 2025 Sep 19. PMID 40970531
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186
- [Derived] Chang FH, Chiu V, Ni P, Lin YN, Kang JH, Liou TH, Lu L, Han DS, Skidmore ER. Enhancing community participation for stroke survivors with cognitive impairment: study protocol for a randomised controlled trial in Taiwan. BMJ Open. 2020 Dec 7;10(12):e040241. doi: 10.1136/bmjopen-2020-040241. PMID 33293312